CLINICAL TRIAL: NCT06297564
Title: Progesterone Primed Endometrial Protocol Versus Gonadotropin-releasing Hormone Antagonist Protocol in Women Undergoing Assisted Reproductive Treatments
Brief Title: Progesterone Primed Endometrial Protocol Versus Gonadotropin-releasing Hormone Antagonist Protocol in Assisted Reproductive Treatments
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Valley University (Other)
Responsible Party: Principal Investigator, Waleed Ahmad Ali, Lecturer of Obstetrics and Gynecology, Faculty of Medicine, New Valley University., New Valley University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07/3/9-2023/4
Record Dates: First submitted 2024-02-22; First posted 2024-03-07 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Progesterone Primed Endometrial Protocol; Gonadotropin Releasing Hormone Antagonist Protocol; Assisted Reproductive Treatments

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progesterone primed endometrial protocol (Active Comparator): The cases were received soft progesterone capsules (brand name: Utrogestan, 100 mg, Laboratories Besins International, France) 100 mg and 150 IU of human menopausal gonadotropin (hMG) concomitantly from the menstrual cycle (MC) day 3 until the trigger day
  Interventions: Other: Progesterone primed endometrial protocol
- Gonadotropin-releasing hormone antagonist protocol (Experimental): The cases were received the gonadotropin-releasing hormone antagonist (GnRH-ant) protocol consisting of HMG 150 IU's daily injection from MC 3 until the trigger day. GnRH-ant (Cetrotide, 0.25 mg, MerckSerono) was started when at least one of the following criteria were met: LH >10 IU/L, the presence of at least one follicle with mean diameter >14 mm, or serum E2 level >600 pg/mL.
  Interventions: Other: Gonadotropin-releasing hormone antagonist protocol

INTERVENTIONS:
Other: Progesterone primed endometrial protocol — The cases were received soft progesterone capsules (brand name: Utrogestan, 100 mg, Laboratories Besins International, France) 100 mg and 150 IU of human menopausal gonadotropin (hMG) concomitantly from the menstrual cycle (MC) day 3 until the trigger day.
  Arms: Progesterone primed endometrial protocol
Other: Gonadotropin-releasing hormone antagonist protocol — The cases were received the gonadotropin-releasing hormone antagonist (GnRH-ant) protocol consisting of HMG 150 IU's daily injection from MC 3 until the trigger day. GnRH-ant (Cetrotide, 0.25 mg, MerckSerono) was started when at least one of the following criteria were met: LH >10 IU/L, the presence of at least one follicle with mean diameter >14 mm, or serum E2 level >600 pg/mL.
  Arms: Gonadotropin-releasing hormone antagonist protocol

SUMMARY:
The aim of this study was to compare the clinical outcomes in progesterone primed endometrial protocol versus gonadotropin-releasing hormone antagonist protocol in women undergoing assisted reproductive treatments.

DETAILED DESCRIPTION:
Utilizing the assisted reproductive techniques (ART) has exhibited a substantial rise within the last years, emerging as a crucial modern medicine component with reliable results.

The utilized protocols for endometrial preparation in ART are aimed at maximizing the treatments' success. Typically, utilizing gonadotropin-stimulating hormone (GnRH) antagonists or agonists remains involved for preventing an early luteinizing hormone (LH) peak along ovulation prior to oocytes retrieval.

The GnRH-antagonist (GnRH-a) protocol is favored by many clinicians as well as patients due to its simplicity, convenience, flexibility, and absence of functional ovarian cysts or "menopausal" symptoms linked to the agonist protocol. Nevertheless, some RCTs' findings address that the antagonist protocol yields a reduced oocytes' number. Additionally, it exhibits lower pregnancy rates as opposed to the agonist extended therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 to 40 years.
* A basal antral follicle count (AFC) <6.
* All patients had to have a body mass index between 18.5 to 29.9 kg/m2.
* Undergoing IVF/ICSI cycles.
* With previous poor response to conventional prolonged therapy utilizing GnRH agonists (retrieving three oocytes).

Exclusion Criteria:

* Cycles with fresh embryo transfer.
* Transfers of cleavage embryos (d2/d3).
* Embryos from cycles with preimplantation genetic screening.
* Cryopreservation of oocytes.
* Oocyte donation cycles.
* Cycles that produced embryos but without et at the time of the analysis.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Women undergoing IVF/ICSI cycles with ages of 21 to 40 years, body mass index between 18.5 to 29.9 kg/m2, with previous poor response to conventional prolonged therapy utilizing GnRH agonists (retrieving three oocytes), along with a basal antral follicle count of less than six. .
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
The number of retrieved oocytes | 34 to 36 hours post HCG administration
  Retrieved oocytes will be collected after ovarian induction by gonadotropin injection

SECONDARY OUTCOMES:
Pregnancy rate | Fourteen days following the transfer
  Biochemical pregnancy was determined as serum HCG higher than 25 mIU/ml at twelve to fourteen days following the transfer. Gynecological ultrasound assessment was accomplished at thirty to thirty-five following the transfer. Additionally, the gestational sac existence was regarded as clinical pregnancy, with the clinical pregnancy rate = (clinical pregnancy cycles' number/ all transfer cycles' number) × 100%. Moreover, live birth rate equals (live birth cycles' number/ all transfer cycles' number) × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- New Valley University, New Valley, New Valley Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.